CLINICAL TRIAL: NCT01737242
Title: UK Genetic Prostate Cancer Study: Epidemiology and Molecular Genetics Studies
Acronym: UKGPCS
Status: Active, not recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 06/MRE02/4; CCR0848
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Prostate Tissue, saliva samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The UKGPCS was set up to find genetic alterations which occur in patients who have prostate cancer.

A man's risk of developing prostate cancer increases if he has a first-degree relative (father or brother) who was diagnosed with prostate cancer at a young age. This is why we are looking for men who are affected at a young age or who have a family history of prostate cancer, since it is more probable that these prostate cancers are due to an inherited genetic cause rather than an environmental cause.

We also ask all men who come to the Royal Marsden Hospital to be treated for prostate cancer if they would like to take part in the study so that we can also look to see if we find genetic alterations in older men, and those who do not have a family history of prostate cancer.

DETAILED DESCRIPTION:
The study is divided into two parts:

1. The Study at The Royal Marsden NHS Foundation Trust, London and Sutton:

   The study will be offered to every patient attending the prostate clinics at The Royal Marsden NHS Foundation Trust, London and Sutton. This is called 'The Systematic Study'.

   Patients are approached in the clinic and are given an information sheet and the study is also explained verbally. They are asked for 18ml of blood and asked to fill out a family history and epidemiological questionnaire. Those who have not had any treatment will also be asked for 18ml blood for serum and plasma marker studies.

   Those patients with one relative affected with PrCa where one is ≤ 65 years at diagnosis or a total of 3 or more relatives with PrCa at any age, will be asked if their relatives can be approached to be asked to give a blood sample for DNA analysis for PrCa predisposition genes and tumour samples for molecular analyses for PrCa predisposition and behaviour as outlined above. Where relatives with PrCa are deceased, pathology records and tumour blocks will be requested after obtaining details of where they were treated via the index case.

   Consent Consent will be sought prospectively from living individuals accrued into the study from January 2006 to access medical records and tumour blocks.

   This study has been active since 1992 and all blood samples have informed consent for PrCa predisposition gene studies. Outside tumour blocks and pathological samples have informed consent for molecular studies. Many of The Royal Marsden NHS Foundation Trust PrCa tumour samples also have consent under a clause in the operation consent form in use at that time that 'material removed may be used for research purposes'. Some tissue was collected from local hospitals under the auspices of the previous protocol and the consent form did not explicitly state separate consent for the use of tissue at that time, although it was part of the approved protocol. Many patients are now deceased. It is therefore proposed that tissue and medical record data collected retrospectively will be analysed anonymously with no results fed back to patients as this would not impact upon their care. An exception is results from the studies on blood where findings in PrCa predisposition genes could have implications for relatives.

   Those patients who are still living who have previously taken part in the study from 1992 until the present and who have not taken part in the environmental questionnaire part of the study will be invited to take part in this part of the study. New consent will be obtained for this.
2. The Study at Collaborative Centres throughout the UK. Many of these are via the NCRN network.

This is conducted as for the Study at The Royal Marsden except the study is explained verbally and then if the patient is interested, their details are given to the study office by confidential fax and the study office sends the patient an information sheet and consent form.

Furthermore, the only groups of patients eligible for this part of the study are (a) men with PrCa presenting at a young age (≤ 60 years) or (b) PrCa in first-degree related pairs where one is ≤ 65 years at diagnosis or (c) a total of 3 or more relatives with PrCa at any age

The two parts (1) and (2) are now called the UKGPCS (UK Genetic Prostate Cancer Study).

There are currently over 300 collaborators UK-wide participating under the auspices of the previous protocol (previously, The Cancer Research UK/British Prostate Group//British Association of Urological Surgeons Section of Oncology and NCRN Familial Prostate Cancer Study).

Proposed analyses on the samples The samples will be used to find PrCa predisposition genes using linkage and other analyses. These investigations are solely for research to find a prostate cancer-predisposing gene and no results would be conveyed to the patients until such a gene(s) had been found. If such a gene(s) is found, then no patient will have genetic testing for abnormalities in such a gene without prior genetic counselling and this would be on a newly taken blood sample. Only those patients who wish (as stated on their consent form) to be informed of research findings will be contacted. If this occurs more than 6 months after the last contact with the patient, this would be via the GP.

Data will be correlated with medical records and treatment outcome to find genetic alterations that are associated with prostate cancer development and/or prognosis.

Tumour material will be collected and stored at -70oC in freezer space currently available at The Institute of Cancer Research. Tumour will also be stored in RNA later and paraffin embedded tumour will be made into tissue microarrays and sections cut. This will be used for molecular biology analysis.

Cases and their relatives may be flagged by the cancer registry to confirm a diagnosis of prostate cancer, a date of death and cause of death. This will be done via the Medical Research Information Service (MRIS), using records maintained by The NHS Information Centre and the NHS Central Register.

Clinical details are collected routinely as part of the medical care and clinical follow up record on patients with prostate cancer and these include disease parameters (e.g. stage, grade) and treatment outcome (e.g. survival data, side effects of treatment). We will also request follow-up data, approximately 2 years after the patient has consented, to record any relapse, treatment and survival data that has occurred since diagnosis. We will link the genetic findings with these clinical data to try to identify genetic markers of disease parameters (e.g. those which predict for poorer prognosis or worse late toxicity from treatments such as radiotherapy). These data would be analysed anonymously after linking the clinical and genetic datasets. No results would be feedback to participants. We will supply anonymised data from this to an EU dataset (Genepi study). This would only be to a central database managed under the auspices of GCP and would only be anonymised data. No individual would be identifiable to the holders of the Genepi database.

ELIGIBILITY:
Inclusion Criteria:

* Man with PrCa at any age at diagnosis at Royal Marsden NHS Foundation Trust
* Those outside the Royal Marsden NHS Foundation Trust with
* PrCa at or below 60 years at diagnosis
* PrCa in first-degree related pairs where one is ≤ 65 years at diagnosis
* PrCa at any age in a cluster with 3 or more cases
* Those able to understand the information sheet and give informed consent (language line is available for those who wish to have translation)
* Any unaffected relatives of men who are already taking part in the study

Exclusion Criteria:

* Man with PrCa who is too ill to take part

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patients that meets the eligibility criteria and may be attending a hospital that have got ethical approval.
Sampling Method: Non-Probability Sample
Enrollment: 23826 (Actual)
Dates: Start 1993-01 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To find genes which predispose to PrCa | 2017

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind A Eeles, FRCP FRCR, Principal Investigator — Institute of Cancer Research and Royal Marsden Hospital
Locations (1):
- Institute of Cancer Research and Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the Data Access Commitee

REFERENCES:
- [Derived] Kote-Jarai Z, Mikropoulos C, Leongamornlert DA, Dadaev T, Tymrakiewicz M, Saunders EJ, Jones M, Jugurnauth-Little S, Govindasami K, Guy M, Hamdy FC, Donovan JL, Neal DE, Lane JA, Dearnaley D, Wilkinson RA, Sawyer EJ, Morgan A, Antoniou AC, Eeles RA; UK Genetic Prostate Cancer Study Collaborators, and the ProtecT Study Group. Prevalence of the HOXB13 G84E germline mutation in British men and correlation with prostate cancer risk, tumour characteristics and clinical outcomes. Ann Oncol. 2015 Apr;26(4):756-761. doi: 10.1093/annonc/mdv004. Epub 2015 Jan 16. PMID 25595936
- See also: Study Website — http://www.icr.ac.uk/ukgpcs